CLINICAL TRIAL: NCT00937196
Title: Effects of Placebos and Verbal Suggestions on Blood Pressure - Randomized Controlled Trial
Brief Title: Placebo Effects on Blood Pressure Induced by Expectancy Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Karin Meissner, PD Dr. med., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KM-DZ-06
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Histaminum hydrochloricum globuli (Active Comparator): To allow double-blind administration of the placebo pills going along with verbal suggestions of a blood-pressure-lowering effect
  Interventions: Drug: Histaminum hydrochloricum globuli
- Placebo globuli (Experimental)
  Interventions: Drug: Placebo globuli
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Placebo globuli — placebo globuli administered together with verbal suggestions of a hypotensive drug effect
  Arms: Placebo globuli
Drug: Histaminum hydrochloricum globuli
  Arms: Histaminum hydrochloricum globuli

SUMMARY:
The objective of the present study was to examine the effects of a single placebo intervention on blood pressure and to investigate autonomic and psychological mediating mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

* not meeting inclusion criteria
* hypotension or hypertension
* treated or untreated hypertension or hypotension
* Severe systemic disorders (tumors, tbc, diabetes, asthma etc)
* diseases that influence the cardiovascular or gastrointestinal system
* intake of drugs affecting blood pressure and/or autonomic nervous system
* pregnancy and lactation phase
* body mass index >= 32
* cardiovascular risk factors (diabetes, smoking)
* drug or alcohol abuse
* insufficient compliance
* participation in another trial within the last three months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure (systolic, diastolic) | minutes 1 to 30 after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karin Meissner, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Institute of Medical Psychology, Ludwig-Maximilians-University Munich, Munich, Germany

REFERENCES:
- See also: Meissner's homepage — http://www.imp.med.uni-muenchen.de/members/mitarbeiter/meissner/index.html